CLINICAL TRIAL: NCT06703229
Title: Assessment of the Impact of Two Dexmedetomidine Dosages Added with Bupivacaine in Ultrasound-Guided Transversus Abdominis Plane Block for Postoperative Analgesia Following Inguinal Hernia Repair: Randomized Controlled Study
Brief Title: Assessment of the Impact of Two Dexmedetomidine Dosages Added with Bupivacaine in Ultrasound-Guided Transversus Abdominis Plane Block for Postoperative Analgesia Following Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Adel Ali Hassan, Lecturer of Anesthesia, Surgical Intensive Care and Pain Management, Faculty of Medicine, Port Said University, Port Said University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT2023-010
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Spinal Anaesthesia; Herniorrhaphy; Transversus Abdominis Plane Block
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group, D1 (Active Comparator): group, D1, had a TAP block that included 0.5 µg/kg of dexmedetomidine and bupivacaine
  Interventions: Drug: The Transversus Abdominis Plane (TAP) block
- group, D2 (Active Comparator): group, D2, received the same block but with 1 µg/kg of dexmedetomidine.
  Interventions: Drug: The transverse abdominis plane (TAP) block

INTERVENTIONS:
Drug: The Transversus Abdominis Plane (TAP) block — or injectate preparation, utilizing ultrasound guidance while the patient was supine. In the D1 group, patients were administered 20 mL of 0.25% isobaric bupivacaine with 0.5 mcg/kg of dexmedetomidine.
  Arms: group, D1
Drug: The transverse abdominis plane (TAP) block — Patients in the D2 group received 20 mL of 0.25% isobaric bupivacaine with 1 mcg/kg of dexmedetomidine.
  Arms: group, D2

SUMMARY:
The principal outcome assessed was the duration until the initial request for analgesia post-surgery. The secondary outcomes encompassed the total quantity of analgesics administered (ketorolac, paracetamol, and morphine) within the initial 24 hours. Pain levels, measured using the Visual Analogue Scale (VAS), were evaluated at rest and during movement at many intervals following surgery (1, 6, 12, and 24 hours). The study also observed postoperative complications, such as emesis, hypotension, bradycardia, and pruritus.

DETAILED DESCRIPTION:
One of the most frequently performed surgical procedures worldwide is the repair of an open inguinal hernia, with a postoperative pain severity of moderate to severe affecting over 60% of patients. Post-surgical analgesia frequently employs a multifaceted approach, incorporating oral pharmacotherapy and regional anesthetic procedures. Opioids are a conventional option for postoperative pain management; nevertheless, their administration is linked to adverse effects such as nausea, vomiting, sleepiness, pruritus, and respiratory depression, which may impede the recovery process. Non-opioid alternatives, however, can improve patient rehabilitation and overall outcomes. The Transversus Abdominis Plane (TAP) block efficiently reduces early postoperative discomfort and decreases narcotic usage, which is a significant advantage for patients undergoing inguinal hernia repair. To alleviate pain in the abdominal wall muscles, peritoneum, and skin, this treatment involves administering a local anesthetic into the space between the transversus abdominis and internal oblique muscles.]2[

ELIGIBILITY:
Inclusion Criteria:

* with ASA physical status I or II
* scheduled for elective unilateral inguinal hernioplasty under spinal anesthesia
* aged 18 to 60 years
* both genders

Exclusion Criteria:

patient refusal, BMI ≥ 40 kg/m2 incapacity to engage in pain assessment contraindications to spinal anesthesia (e.g., coagulopathy, skin infection)

- and intolerance to the research medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
the initial request for analgesia post-surgery | 24 hours
  The postoperative Visual Analogue Scale (VAS) is a 10 cm horizontal line labeled "no pain" at one end and "worst pain" on the other end.

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian liver hospital, Al Mansurah, Ansoura, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.